CLINICAL TRIAL: NCT00209651
Title: Phase II Study of Oral S-1 Plus Irinotecan in Patients With Advanced Colorectal Cancer: Hokkaido Gastrointestinal Cancer Study Group HGCSG0302
Brief Title: Phase II Study of Oral S-1 Plus Irinotecan (IRIS) in Patients With Advanced Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hokkaido Gastrointestinal Cancer Study Group (Other)
Collaborators: Hokkaido University Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HGCSG0302; IRIS
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2007-11-01 (Estimated); Status verified 2007-10

CONDITIONS: Colorectal Cancer
Keywords: Irinotecan, S-1, Phase II, colorectal cancer,
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Irinotecan; titanium silicide; S 1 (combination)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Irinotecan and S-1
  Interventions: Drug: Campto, Topotesin; Drug: TS-1

INTERVENTIONS:
Drug: Campto, Topotesin — q00 mg/m2, IV (in the vein) on day 1,15 of each 28 day cycle.
  Other Names: irinotecan
Drug: TS-1 — 80 mg/m2, PO (oral) on day 1~14 of each 28 day cycle.
  Other Names: S-1

SUMMARY:
To assess the usefulness of irinotecan plus S-1 therapy based on the antitumor effect and survival period. by performing a phase II study of this combination in patients with inoperable or with postoperative colorectal cancer.

DETAILED DESCRIPTION:
A multicenter Open-label, single-arm, phase II clinical trial is conducted on patients with histological stage IV colorectal cancer given irinotecan plus S-1. The usefulness of this regimens as 1st line therapy for colorectal cancer was evaluated by the disease-free survival rate (DFR), overall survival rate (OS), incidence and severity of adverse event.

ELIGIBILITY:
Inclusion Criteria:

1. Histological diagnosis of colorectal adenocarcinoma.
2. Measurable or assessable lesions.
3. Age: 18 ~ 75 years.
4. Performance Status (ECOG): 0 ~ 2.
5. No prior chemotherapy or only one regimen of previous chemotherapy (with a washout period >4 weeks after the final day of the previous therapy). Adjuvant chemotherapy is not defined as previous therapy.
6. No history of treatment with CPT-11 or S-1.
7. No history of radiotherapy to the abdomen.
8. Oral intake of S-1 is possible.
9. Adequate function of major organs (bone marrow, heart, lungs, liver etc.). WBC 3,500/mm3 and 12,000/mm3. Hb 10.0 g/dl. Platelet count 100,000/mm3. GOT and GPT 2.5times the upper limit of normal (excluding liver metastasis). T-Bil 2.0mg/dl. Creatinine <1.5 mg/dl (but if it is 1.0 ~ 1.5 mg/dl, the dose of S-1 can be decreased according to the dose reduction criteria to allow registration in the trial). Normal ECG (not considering clinically unimportant arrhythmias and ischemic changes).
10. Predicted survival for >3 months.
11. Able to give written informed consent

Exclusion Criteria:

1. Severe pleural effusion or ascites.
2. Metastasis to the central nervous system (CNS).
3. Active gastrointestinal bleeding.
4. Active infection.
5. Diarrhea (watery stools).
6. Uncontrolled ischemic heart disease.
7. Serious complications (such as intestinal paralysis, intestinal obstruction, interstitial pneumonia or pulmonary fibrosis, uncontrolled diabetes mellitus, heart failure, renal failure, or hepatic failure).
8. Active multiple cancer.
9. Severe mental disorder.
10. Pregnancy, possible pregnancy, or breast-feeding.
11. Flucytosine treatment
12. Gilbert's syndrome (4).
13. Judged to be ineligible for this protocol by the attending physician.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2004-01; Study Completion 2007-12 (Estimated)

PRIMARY OUTCOMES:
objective tumor response | 1-year

SECONDARY OUTCOMES:
Response duration, time to progression, overall survival, and safety will also be assessed. | 2-years

CONTACTS AND LOCATIONS:
Overall Officials: Yoshito Komatsu, MD.PhD, Study Chair — Hokkaido Gastrointestinal Cancer Study Group
Locations (1):
- Hokkaido University Hospital, Sapporo, Hokkaido, Japan